CLINICAL TRIAL: NCT07329153
Title: Neuronavigated and Non-Neuronavigated Accelerated Intermittent Theta-Burst Stimulation for Treatment-Resistant Depression A Sham-Controlled Randomized Controlled Trial
Brief Title: Neuronavigated aiTBS for TRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of California, San Diego (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Andre Russowsky Brunoni, Professor and Chief of the Division of Interventional Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2025-1926
Record Dates: First submitted 2026-01-07; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression (TRD)
Keywords: depression; TMS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Neuronavigated aiTBS (Experimental): TBS device placement during treatment determined by MRI imaging
  Interventions: Device: aiTBS
- Non-Neuronavigated aiTBS (Active Comparator): Conventional device placement during treatment
  Interventions: Device: aiTBS
- Sham aiTBS (Sham Comparator): identical procedures as the other 2 groups but without turning on the device
  Interventions: Device: aiTBS

INTERVENTIONS:
Device: aiTBS — Repetitive transcranial magnetic stimulation (rTMS) interventions - accelerated intermittent theta-burst stimulation (aiTBS) and individualized neuronavigation.

SUMMARY:
The purpose of this study is to confirm the efficacy of two recently introduced repetitive transcranial magnetic stimulation (rTMS) interventions - accelerated intermittent theta-burst stimulation (aiTBS) and individualized neuronavigation - in treatment-resistant depression (TRD). Using a three-arm design (neuronavigated aiTBS, non-neuronavigated aiTBS, and sham), this randomized controlled trial (RCT) is the first to specifically investigate the incremental benefit of neuronavigation within an accelerated stimulation protocol, as well as the first confirmatory RCT comparing the efficacy of each of these active treatments vs. sham, overcoming previous generalizability issues and being conducted in an independent, multicenter US TRD sample.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years at the time of consent
2. Diagnosis: Current major depressive episode (MDE) in the context of unipolar major depressive disorder (MDD), as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), confirmed by clinical psychiatric interview
3. Treatment Resistance: Documented failure to respond to at least two adequate antidepressant trials on the Antidepressant Treatment History Form-Short Form (ATHF-SF). An adequate trial is defined as:

   1. Antidepressant medication at the maximum tolerated dose for at least 6 weeks, OR
   2. Evidence-based psychotherapy consisting of at least 12 sessions
4. Depression Severity: Montgomery-Åsberg Depression Rating Scale (MADRS) score >19 at screening, indicating moderate to severe depression
5. Medication Stability: No changes in antidepressant medication type or dose for at least 6 weeks prior to randomization. Stable doses of permitted medications must be maintained throughout the trial
6. Informed Consent: Demonstrated capacity to provide written informed consent and comply with study procedures
7. Availability: Ability to attend treatment sessions for 15 consecutive workdays (approximately 90 minutes per day) and complete assessments including 4-hour evaluations at baseline and endpoint

Exclusion Criteria:

Psychiatric Exclusions:

1. Any psychiatric disorder other than MDD and comorbid anxiety disorders, including but not limited to:

   (i) Bipolar disorder (Type I or II) (ii) Schizophrenia spectrum or other psychotic disorders (iii) Post-traumatic stress disorder (PTSD) (iv) Attention-deficit/hyperactivity disorder (ADHD) (v) Autism spectrum disorder (ASD) (vi) Obsessive-compulsive disorder (OCD) (vii) Current DSM-5 substance-use disorder (abuse or dependence) within the past 6 months, except nicotine dependence
2. Personality disorder confirmed on clinical interview by an experienced study psychiatrist
3. Severe suicidal ideation with structured plan (HDRS-17 item 3 score >2) or as determined by the evaluating psychiatrist
4. Depressive symptoms better explained by another psychiatric condition, a medical condition, substance use, or use of medications

Medical and Neurological Exclusions:

1. Any neurological disorder including but not limited to:

   (i) History of seizure disorder or epilepsy (ii) Family history of epilepsy (first-degree relatives) (iii) Significant head trauma with loss of consciousness >5 minutes (iv) Stroke or transient ischemic attack (v) Neurodegenerative disorders (e.g., Parkinson's disease, multiple sclerosis, dementia) (vi) Brain tumor or intracranial mass lesion
2. Unstable medical condition, defined as any condition requiring acute medical intervention or hospitalization within the past 3 months, or any condition that in the investigator's judgment could affect participant safety or study outcomes

Contraindications to TMS/MRI:

1. Presence of ferromagnetic material in or near the head, including:

   (i) Intracranial implants (e.g., aneurysm clips, shunts, stimulators) (ii) Cochlear implants or hearing aids (iii) Metallic facial tattoos or permanent makeup (iv) Other implanted medical devices deemed unsafe for MRI/TMS
2. Inability to tolerate MRI scanning due to claustrophobia or other reasons

Medication Exclusions:

Current use of medications known to significantly alter cortical excitability:

1. Anticonvulsants (including those used for mood stabilization)
2. Psychostimulants
3. Lithium
4. Benzodiazepines exceeding 10mg diazepam-equivalent daily dose

Prior Treatment Exclusions:

1. Electroconvulsive therapy (ECT) (≥ 6 sessions) in the current depressive episode
2. Ketamine or esketamine treatment (≥ 6 sessions) in the current depressive episode
3. Use of rTMS/iTBS (≥ 15 sessions) during the current depressive episode
4. Vagus nerve stimulation (VNS) or deep brain stimulation (DBS) implantation

Psychotherapy:

• Concurrent evidence-based psychotherapy is permitted if initiated >4 weeks prior to enrollment and maintained at stable frequency throughout the tria

Other reasons:

1. Unable to adhere to the study visit schedule
2. Planning to relocate outside the study catchment area during the trial period
3. No reliable transportation to attend study visits
4. Current participation in another research study
5. Current pregnancy (confirmed by in interview and clinical evaluation and, if deemed necessary, urine pregnancy test at screening)
6. Currently breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2031-06 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
HDRS-17 - Depression severity assessment | From Baseline visit until week 5 visit
  depression severity as assessed by the Hamilton Depression Rating Scale-17 items (HDRS-17)

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | From Baseline visit until week 5 visit.
Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR) | From Baseline visit until week 5 visit
  participant self-rated symptomatology

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California at San Diego (UCSD), San Diego, California
  - Cornell University, New York, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas